CLINICAL TRIAL: NCT06220864
Title: A Phase 1, Open-Label Dose Escalation and Expansion Study of SNV1521 in Participants with Advanced Solid Tumors
Brief Title: SNV1521 in Participants with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Synnovation Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNV1521-101
Record Dates: First submitted 2024-01-12; First posted 2024-01-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose Escalation (Experimental)
  Interventions: Drug: SNV1521
- Dose Expansion (Experimental)
  Interventions: Drug: SNV1521
- Combination Dose Escalation (Experimental)
  Interventions: Drug: SNV1521; Drug: Trastuzumab Deruxtecan
- Dose Expansion for Metastatic Castration Resistant Prostate Cancer (Experimental)
  Interventions: Drug: SNV1521
- Dose Expansion for Pancreatic Ductal Adenocarcinoma (Experimental)
  Interventions: Drug: SNV1521
- Dose Expansion for Solid Tumors with Brain Metastases (Experimental)
  Interventions: Drug: SNV1521

INTERVENTIONS:
Drug: SNV1521 — SNV1521 is a tablet taken orally. Dose and frequency are dependent upon treatment arm.
Drug: Trastuzumab Deruxtecan — Trastuzumab Deruxtecan is given as an infusion based upon prescribing information.
  Arms: Combination Dose Escalation

SUMMARY:
This study is testing a new medicine, SNV1521, for people with advanced cancers. The researchers want to find out if SNV1521 is safe, well-tolerated, and effective in treating solid tumors. They are investigating different doses in order to find the most effective and safe one. They are also investigating whether it can be combined with other cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic solid tumor malignancy
* Evaluable or Measurable disease (RECIST 1.1 Criteria).
* ECOG Performance Status 0 or 1.
* Life expectancy > 3 months

Exclusion Criteria:

* History of other malignancy within the past 2 years
* Prior diagnosis of Myelodysplastic syndrome or Acute Myeloid Leukemia
* Significant cardiovascular disease within 6 months
* Significant gastrointestinal disease
* HIV infection with a CD4+ T-cell count < 200 cells/μL and/or a detectable viral load
* Liver dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety of SNV1521 | From first dose through last dose (up to 13 months)
  Treatment emergent adverse events (TEAEs)
Tolerability of SNV1521 | DLTs: From first dose through completion of first cycle (28 days)
  Incidence and frequency of dose-limiting toxicities (DLTs) (Dose-escalation arm only)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Yale University, New Haven, Connecticut
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - START Center for Cancer Care, West Valley City, Utah
- Australia (4):
  - Scientia Clinical Research, Randwick, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Crawley, Western Australia